CLINICAL TRIAL: NCT07324759
Title: Effect of Saffron Extract Capsule Supplement on Skin Rejuvenation and Anti-Ageing in Healthy Adult Male and Female Subjects: Randomised, Double-Blind, Two-Group, Prospective, Multi-Centre Exploratory Study
Brief Title: Clinical Study to Assess Safety, Effectiveness and In-Use Tolerability of Saffron Extract Capsules for Improving Skin Health and Reducing Signs of Aging on Healthy Adult Male and Female Subjects.
Acronym: GLOW
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Pharmanza Herbal Private Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NB250038-PH_1.0_20Dec25
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Wrinkles; Fine Lines; Hyperpigmentation; Dark Spots
MeSH Terms: conditions — Hyperpigmentation | interventions — Calcium Carbonate; 6-hydroxy-5-((p- sulfophenyl)azo)-2-naphthalenesulfonic acid disodium salt; Starch; Talc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized Saffron Extract (Crocus Sativus L) 10 mg Capsule (Experimental): Mode of Usage: Administer one capsule once daily after meal, ideally at the same time each day to maintain consistency in absorption. Swallow the capsule whole with a full glass of water; do not crush, break, or chew the capsule.
  Frequency: Once a day, after lunch Route of administration: Oral Storage Condition: Store in cool and dry place, away from sunlight, heat and moisture.
  Interventions: Dietary Supplement: Standardized Saffron Extract (Crocus Sativus L) 10 mg Capsule
- Placebo ( Maltodextrin, Calcium carbonate, Sunset yellow, Maize starch, Mg Stearate, Talc) (Placebo Comparator): Mode of Usage: Administer one capsule once daily after meal, ideally at the same time each day to maintain consistency in absorption. Swallow the capsule whole with a full glass of water; do not crush, break, or chew the capsule.
  Frequency: Once a day, after lunch Route of administration: Oral Storage Condition: Store in cool and dry place, away from sunlight, heat and moisture.
  Interventions: Other: Placebo (capsules containing Maltodextrin, Calcium carbonate, Sunset yellow, Maize starch, Mg Stearate, Talc)

INTERVENTIONS:
Dietary Supplement: Standardized Saffron Extract (Crocus Sativus L) 10 mg Capsule — Mode of Usage: Administer one capsule once daily after meal, ideally at the same time each day to maintain consistency in absorption. Swallow the capsule whole with a full glass of water; do not crush, break, or chew the capsule.
  Frequency: Once a day, after lunch Route of administration: Oral Storage Condition: Store in cool and dry place, away from sunlight, heat and moisture.
  Arms: Standardized Saffron Extract (Crocus Sativus L) 10 mg Capsule
Other: Placebo (capsules containing Maltodextrin, Calcium carbonate, Sunset yellow, Maize starch, Mg Stearate, Talc) — Mode of Usage: Administer one capsule once daily after meal, ideally at the same time each day to maintain consistency in absorption. Swallow the capsule whole with a full glass of water; do not crush, break, or chew the capsule.
  Frequency: Once a day, after lunch Route of administration: Oral Storage Condition: Store in cool and dry place, away from sunlight, heat and moisture.
  Arms: Placebo ( Maltodextrin, Calcium carbonate, Sunset yellow, Maize starch, Mg Stearate, Talc)

SUMMARY:
This is a randomized, double-blind, comparative, two-arm, prospective, interventional, multi-centre clinical study to evaluate the safety, efficacy, and in-use tolerability of test products, standardized saffron extract capsules, on skin rejuvenation and age-defying benefits in healthy adult male and female subjects.

DETAILED DESCRIPTION:
A total of 50 male and non-pregnant, non-lactating female subjects aged 30-55 years will be enrolled, with 25 subjects assigned to each product group (Test Product A and B). Approximately 40 subjects in total (20 per group) are expected to complete the study.

Subjects will be randomized in a 1:1 ratio to receive either one of the two test treatments: 25 subjects in Test Product A and 25 subjects in Test Product B and 40 subjects will complete the study (20 subjects/treatment).

The potential subjects will be screened as per the inclusion and exclusion criteria only after obtaining written informed consent from the subjects. Subjects will be contacted telephonically by recruiting department prior to the screening.

There will be total of 5 visits during the study. The duration of the study will be 120 Days (16 weeks) from the enrolment. Subjects will be instructed to visit the facility as per below visits:

* Visit 01 (Day 07 days prior to Day 01): Screening, ICD obtained, Medical history, Sleep Diary, Safety laboratory parameters
* Visit: 02 (Day 01, Week 00): Enrolment, Baseline assessments.
* Visit 03 (Day 45, Week 06): Product Phase, Evaluations
* Visit 04 (Day 90, Week 12): Evaluations, Safety laboratory parameters and End of Product Phase
* Visit 05 (Day 120, Week 16): Instrument Evaluations only and End of Study

ELIGIBILITY:
Inclusion Criteria:

1. Age: 30 to 55 years (both inclusive) at the time of consent.
2. Sex: Adult male and female having wrinkles and fine lines at crow feet's area, facial hyperpigmentation and dark spots such as tan, pimple marks, sunspots, age spots, uneven skin tone on both side of face.
3. Females of childbearing potential should have a self-reported negative urine pregnancy test at the time of screening visit.
4. Subjects should not have used any cosmetic, nutraceutical or therapeutic products for skin ageing in last 1 month.
5. Subjects must be willing to stop using any cosmetics or any medical products for skin ageing for the duration of the study.
6. Subjects are not allowed to participate in any other study until this study is complete.
7. Subjects must be willing and able to follow the study directions and to return for all specified visits with the product.
8. Subjects must agree to record each use of the test products in the subject's diary card on daily basis.
9. Subjects must agree to record medication use during the study.

Exclusion Criteria:

1. Subjects who are on steroids for last six months and using immunosuppressive, anti-inflammatory, or hormone-modulating medications that may interfere with study outcomes.
2. Subjects who have used any cosmetic, nutraceutical or therapeutic products for skin last one months.
3. Subjects currently using any oral supplement and topical products containing kojic acid, glycolic acid, niacinamide, alpha arbutin, vitamin C, retinoids, peptides, exfoliating acids, or any other skin-lightening, anti-ageing, or depigmenting agents within the past 4 weeks.
4. Subjects with a known history of hypersensitivity, allergic reactions, or intolerance (such as drowsiness, stomach discomfort, nausea, or vomiting).
5. Subjects with other dermatologic diseases whose presence or products could interfere with the assessment of study.
6. Subjects that are pregnant and/or breastfeeding.
7. The subject has a known allergy or sensitivity to product ingredients.
8. Subjects if do not agree to limit sun exposure to affected areas such as face during prolonged sun exposure.
9. The subject has any other skin conditions i.e. cuts, scratches, ring worms, etc. which in the opinion of the Investigator, will interfere with the study results or will create undue risk for the subject.
10. The subject has any of the conditions or factors that the Investigator believes may affect the response of the skin or the interpretation of the test results.
11. The subject is currently taking or has taken any medication, which the Investigator believes may influence the interpretation of the data.
12. Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of test products in terms of change in facial wrinkles and finelines of Crow's feet area, skin texture -dryness, roughness, smoothness, pores within and between product groups | Baseline on Day 01 and post usage of test products on Day 45 (±2 Days), Day 90 (±2 Days), Day 120 (±2 Days)
  By using Visioscan® VC 20 Plus
To evaluate the effectiveness of test products by assessing change in skin tone - L*, a*, b*, and ITA within and between product groups | Baseline on Day 01 and post usage of test products on Day 45 (±2 Days), Day 90 (±2 Days), Day 120 (±2 Days)
  By using Skin Colorimeter CL 400

SECONDARY OUTCOMES:
To evaluate the effectiveness of test products by assessing change in skin elasticity and firmness within and between product groups | Baseline on Day 01 and post usage of test products on Day 45 (±2 Days), Day 90 (±2 Days), Day 120 (±2 Days)
  By using Cutometer Dual MPA 580 (R0 and R2)
To evaluate the effectiveness of test products by assessing change in skin texture such as skin dryness, redness, fine lines, coarse wrinkles, laxity, roughness and sallowness within and between product groups | from baseline on Day 01 and post usage of test products on Day 45 (±2 Days) and Day 90 (±2 Days)
  By Physician Global Assessment (PGA) using Griffith's scale by Dermatologist or dermatologist trained evaluator
To evaluate the effectiveness of test products by assessing change in wrinkles within and between product groups | from baseline on Day 01 and post usage of test products on Day 45 (±2 Days) and Day 90 (±2 Days)
  Evaluated through Dermatological Evaluation using Glogau Scoring Scale
4. To evaluate the effectiveness of test products by assessing change in skin pigmentation evaluated through Dermatological Evaluation using Skin Pigmentation Scoring within and between product groups. | From baseline on Day 01 and post usage of test products on Day 45 (±2 Days) and Day 90 (±2 Days)
  By using Melasma Area and Severity Index Scale
To evaluate the effectiveness of test products by assessing change in skin hydration within and between product groups | Baseline on Day 01 and post usage of test products on Day 45 (±2 Days), Day 90 (±2 Days), Day 120 (±2 Days)
  Using Corneometer® CM 825
To evaluate the effectiveness of test products by assessing change in skin thickness and density (Skin Ultrasound) within and between product groups. | Baseline on Day 01 and post usage of test products on Day 90 (±2 Days)
  Using Mindray DC 70 or similar
To evaluate the effectiveness of test products by assessing change in visual appearance of facial skin within and between product groups. | baseline on Day 01 and post usage of test products on Day 45 (±2 Days), Day 90 (±2 Days), Day 120 (±2 Days)
  By using Visioface® RD
To evaluate the effectiveness of test products by assessing change in Blood Biomarkers within and between product groups | From baseline on Day 01 and post usage of test products on Day 90 (±2 Days)
  Malondialdehyde, Total Antioxidant Capacity, Glutathione Levels, Procollagen Type-I C-Peptide, Filaggrin, Salivary Cortisol, Lysozyme Levels
To evaluate the effectiveness of test products by assessing change in sleep pattern by mood and sleep diary within and between product groups. | From baseline (Days -07) and Day 90 for Basic Nordic Sleep Questionnaire and PROMIS Sleep Disturbance and Distress Scale baseline (Day -07), Day 01 and post usage of test products on Day 45 (±2 Days), Day 90 (±2 Days), Day 120 (±2 Days)
  evaluated using Basic Nordic Sleep Questionnaire and PROMIS Sleep Disturbance and Distress Scale
To evaluate the effectiveness of test products by assessing change in hair thickness and density within and between product groups | baseline on Day 01 and post usage of test products on Day 45 (±2 Days), Day 90 (±2 Days), Day 120 (±2 Days)
  Using CASLite Nova
To evaluate the effectiveness of the test products by assessing change in stress level within and between product groups. | From baseline on Day 01 and post usage of test products on Day 45 (±2 Days) and Day 90 (±2 Days)
  Using World Health Organization - Quality of Life Questionnaire-BREF
To evaluate the effectiveness of test products by assessing change in general skin condition - lines/ wrinkles, age spots, elasticity/firmness, smoothness, radiance, tone within and between product groups. | From baseline on Day 01 and post usage of test products on Day 45 (±2 Days), Day 90 (±2 Days) and 120 (±2 Days)
  Using Visual Analogue Scale (VAS) score
To evaluate the effectiveness of test products by assessing changes in quality of life regarding test treatment's effect on daily life activities within and between product groups. | Baseline on Day 01 and post usage of test product on Day 45 (±2 Days), Day 90 (±2 Days), Day 120 (±2 Days)
  Using Dermatology Life Quality Index (DLQI)

OTHER OUTCOMES:
To evaluate the safety of the test product by clinical laboratory parameters | From baseline on 07 days prior to day 01 to post-product on Day 90 (±2 Days).
  complete blood count (CBC), Biochemistry, Urinalysis
To evaluate the safety of the test product | Post-product on Day 45(±2 Days) and Day 90 (±2 Days)
  By the monitoring of product emergent systematic evaluation of adverse events
To evaluate the safety of the test treatment by checking compliance towards the test treatments and daily diary entries | From baseline to post-treatment on Day 45(±2 Days) and Day 90 (±2 Days)
  For compliance-capsule counts

CONTACTS AND LOCATIONS:
Overall Officials: Nayan Patel, Principal Investigator — NovoBliss Research Pvt Ltd